CLINICAL TRIAL: NCT05748236
Title: The Efficacy and Safety of Lamotrigine Versus Carbamazepine in Focal Epilepsy: A Randomized, Open Label Clinical Trial in Dhaka Medical College Hospital
Brief Title: The Efficacy and Safety of Lamotrigine Versus Carbamazepine in Focal Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Dhaka Medical College (Other)
Responsible Party: Principal Investigator, Dr. Reaz Mahmud, Assistant Professor, Dhaka Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERC-DMC/ECC/2022/330
Record Dates: First submitted 2023-02-07; First posted 2023-02-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Focal Epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — Lamotrigine; Carbamazepine; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lamotrigine (Active Comparator): Starting dose 25mg once daily for 2 weeks, then 50 mg once daily for next 2 weeks . Then dose will be increased until seizure control or side effects develop (Maximum 500 mg/day)
  Interventions: Drug: Lamotrigine tablet
- Carbamazepine (Active Comparator): Starting dose 100mg twice daily for 2 weeks, then 200 mg twice daily for next 2 weeks. Then dose will be increased until seizure control or side effects develop (Maximum 1600 mg/day)
  Interventions: Drug: Carbamazepine-Containing Product in Oral Dose Form

INTERVENTIONS:
Drug: Lamotrigine tablet — Lamotrigine: Starting dose 25mg once daily for 2 weeks, then 50 mg once daily for next 2 weeks . Then dose will be increased until seizure control or side effects develop (Maximum 500 mg/day).
  Other Names: Lamitrin, Lamogin
  Arms: Lamotrigine
Drug: Carbamazepine-Containing Product in Oral Dose Form — Starting dose 100mg twice daily for 2 weeks, then 200 mg twice daily for next 2 weeks. Then dose will be increased until seizure control or side effects develop (Maximum 1600 mg/day).
  Other Names: Tegretol
  Arms: Carbamazepine

SUMMARY:
Epilepsy is a serious chronic brain disorder that has a tendency towards recurrent seizures. This affects millions of people throughout the world and brings a heavy socioeconomic burden. The treatment of focal epilepsy is more challenging. Selecting an appropriate antiepileptic drug (AED) remains difficult because the chosen drug must be effective, safe and tolerable. It is important to consider the safety and efficacy of an AED for monotherapy separately. The goal of AED therapy is to achieve seizure control with little or no adverse efects, improve the patient's quality of life and ensure patient satisfaction. Different AEDs can be used to treat focal seizures in adults. First line medication for treating focal seizures is carbamazepine (CBZ), but it has drawbacks such as adverse effects including Steven Johnson syndrome, drug interactions and blood dyscrasia. There is also genetic linkage that Steven-Johnson syndrome and toxic epidermal necrolysis with carbamazepine are more common in individuals of Asian descent who carry the HLA-B 1502 allele. Another 1st line drug is lamotrigine (LTG) , it has favourable side effect profile including less sedative effect, less cognitive impairment, less drug interactions and blood dyscrasia. It has an elimination half- life longer than 24 hour, so once daily dosing is possible and it is associated with good drug compliance. Because of its favorable pharmacokinetics and side effect profile, LTG may be preferred to CBZ for focal epileptic seizures. In a study showed that the seizure freedom rate at the end of 6 months was 65% in LTG group compared to 73% in CBZ group. 41% in CBZ group and 32% in LTG group had at least one adverse effects.

Few trials have compared the effectiveness and safety of LTG with CBZ as monotherapy for focal seizures worldwide. By far, no study has yet been conducted addressing the issue of efficacy and safety between lamotrigine and carbamazepine among focal epilepsy patients in the context of Bangladeshi population. Since the usage of LTG is less common in Bangladesh, comparative study of efficacy and safety of LTG versus CBZ will be expected to give more confidence for the use of the drug. Considering this, the study aims to assess the safety and efficacy of carbamazepine and lamotrigine among focal epilepsy patients. This study finding have an implication in the treatment protocol which will be beneficial for the patients and physicians as well.

DETAILED DESCRIPTION:
This prospective hospital based open label interventional study will be conducted in Dhaka Medical College Hospital, Dhaka after receiving approval of this protocol from ethical review committee of DMC. Patients who match the inclusion and exclusion criteria will be enrolled in the study by simple random sampling. A written informed consent will be taken from patients or from their legal attendants after describing the aim, purpose and procedure of the study. Focal epilepsy will be diagnosed according to the criteria of the Commission on Classification and Terminology of the International League against Epilepsy (2017). In this study patients will be divided into 2 groups on their antiepileptic medication. The screening procedure, randomization and drugs will be started at day 1. All the assessment will be completed at day 1 and will be considered as baseline. Randomization will be done at 1:1 into parallel group. Each group will include 34 patients. Group A will include focal epileptic patients on lamotrigine and group B will include focal epileptic patients on carbamazepine. A structured questionnaire will be completed by investigator from answers of participating patients or with the help of their legal attendants, to obtain information on demographic characteristics (age, gender, marital status, education, socioeconomic level etc) and outcome of drug intervention. The patients will maintain a diary during the whole period and ask to note down any seizure frequency with date, time, duration and adverse effects of drugs. During the data record keeping every patient will be evaluated initially by investigator and later independently evaluated by a consultant neurologist.

Lamotrigine will be given at starting dose 25 mg once daily for 2 weeks, then 50 mg once daily for next 2 weeks and carbamazepine will be given at starting dose 100 mg twice daily for 2 weeks, then 200 mg twice daily for next 2 weeks. In both drugs dose will be increased until seizure control or side effects develop.

Patients will be followed up at 1st month, 3rd month and 6th month after receiving medication and following outcome will be assessed: reduction of seizure frequency, seizure free period, hospital readmission, frequency of status epilepticus, all-cause mortality, adverse drug reactions. Patients will be followed up at epilepsy clinic / outpatient department (OPD) and those patients who fail to attend at epilepsy clinic / OPD, by telephonic interview. All the above information will be recorded in a data collection form consisting of relevant questionnaire. After completion, data analysis will be done by SPSS version 26 (Chicago, Illinois, USA).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years regardless of gender.
* Newly diagnosed focal epilepsy patient with or without secondary generalization.
* Relapse following antiepileptic drug withdrawal or failure on treatment other than lamotrigine or carbamazepine.
* Willing to participate and give informed written consent.

Exclusion Criteria:

* Patient with generalized seizure.
* Cryptogenic or unknown onset seizure.
* Known hypersensitivity to medication.
* History of drug abuse.
* Patient with serious medical conditions such as cardiovascular diseases, hepatic failure, renal failure, malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The efficacy and safety between lamotrigine and carbamazepine among focal epilepsy patients. | 6 month
  The measurement of a medicine desired effect under ideal conditions, such as clinical trial (European medicine agency). It is measured as treatment retention rate at the end of follow up and percentage in reduction of seizure frequency from the time of drug initiation

SECONDARY OUTCOMES:
Reduction of seizure frequency. | 6 month
  The frequency of seizure was calculated as the number of seizure events before initial visit and at every follow up visit. The difference of seizure frequency was calculated by subtracting number of events from the previous value. In epilepsy clinic patients are asked to maintain a diary of seizure events with date, time and duration which are kept written in patient record form.
Duration of seizure free period. | 6 month
  It will be evaluated as percentage of patients who are seizure free at the end of follow up period.
Hospital readmission after receiving intervention | 6 month
  In previously admitted patient, is there any readmission?
Rate of death among patients | 6 month
  Death during study period
Adverse drug reactions among two groups. | 6 month
  Any noxious, unintended and undesired effect (including an abnormal laboratory finding) of a drug which occurs at a dose used in humans for prophylactic, diagnostic or therapeutic purpose (WHO).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mohammad Osman, MBBS, Principal Investigator — MD Neurology Thesis; Kazi Gias Uddin Ahmed, MD, Study Chair — Associate professor, Dhaka Medical College; Reaz mahmud, Study Director — Dhaka Medical College
Locations (1):
- Dhaka medical college, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
demographic variables, primary and secondary outcomes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: october 2023 to september 2024
Access Criteria: who work with focal epilepsy patients